CLINICAL TRIAL: NCT06122493
Title: Optimization of Treatment Strategy for Unresectable cN3 Esophageal Squamous Cell Carcinoma: a Phase Ⅱ Single Arm Prospective Study
Brief Title: Optimization of Treatment Strategy for Unresectable cN3 Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RuijinH 2022(270)
Record Dates: First submitted 2023-10-18; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: ESCC; cN3; radiotherapy; chemotherapy; immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — spartalizumab; Taxes; Carboplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Chemotherapy includes carboplatin (AUC = 5, d1) and nab-paclitaxel (175 mg/m², day1) every 3 weeks for four cycles. Simultaneously, immunotherapy with tislelizumab (200 mg) is integrated into the treatment plan for these cycles. After the initial four cycles, patients have physical exams and imaging. Those with SD, PR, or CR receive radiotherapy targeting esophageal lesions and positive lymph nodes, with a total dose of 50.4 Gy over 28 fractions. During radiotherapy, two additional cycles of immunotherapy with tislelizumab are given at three-week intervals. After radiotherapy, patients continue with maintenance treatment, taking tislelizumab every three weeks. This maintenance therapy lasts up to a year, or until disease progression or intolerance develops.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy-immunotherapy-radiotherapy (Other): Carboplatin (AUC = 5, d1) and nab-paclitaxel (175 mg/m², day1) will be administered every 3 weeks for four cycles.Tislelizumab (200 mg) will be administered every 3 weeks for up to 12 months. Radiotherapy targeting esophageal lesions and positive lymph nodes, with a total dose of 50.4 Gy over 28 fractions will be delivered.
  Interventions: Drug: Tirelizumab; Drug: Nab paclitaxel; Drug: Carboplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Tirelizumab — immunotherapy, 200 mg on day 1 per 3 weeks
  Other Names: anti-PD-1 monoclonal antibody
Drug: Nab paclitaxel — chemotherapy, 175 mg/m² on day 1 per 3 weeks
  Other Names: Chemotherapy drug
Drug: Carboplatin — chemotherapy, AUC=5 on day 1 per 3 weeks
  Other Names: Chemotherapy drug
Radiation: Radiotherapy — Patients without disease progression after four cycles of chemoimmunotherapy receive radiotherapy targeting esophageal lesions and positive lymph nodes, with a total dose of 50.4 Gy delivered over 28 fractions.
  Other Names: Locoregional therapy

SUMMARY:
This study aims to investigate a comprehensive therapeutic approach for patients with unresectable esophageal squamous cell carcinoma, clinically staged as Tany, N3, M0, and who are not candidate for concurrent chemoradiotherapy combined with immunotherapy. The approach entails combining chemotherapy with immune therapy, followed by synchronized radiotherapy during the immune maintenance phase. The primary goal is to mitigate treatment-related side effects and enhance the overall prognosis through the integration of these treatment modalities.

DETAILED DESCRIPTION:
Eligible ESCC patients receive a four-cycle regimen of combined chemotherapy plus immunotherapy. Those without disease progression then get definitive radiotherapy with immune maintenance therapy for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal squamous cell carcinoma confirmed through histopathology.
* Distant metastasis excluded by CT, MRI, or PET/CT examinations.
* Locally advanced stage: AJCC/UICC eighth edition staging with any T, N3M0.
* Expected survival time of at least 6 months.
* With an ECOG performance status of 0 to 2. Not accompanied by severe pulmonary hypertension, cardiovascular disease, peripheral vascular disease, severe chronic heart disease, or other comorbidities that could impact radiotherapy progress.
* Adequate function of major organs: Hematopoietic function: Hemoglobin ≥100g/L, platelets ≥90×109/L, white blood cells ≥4×109/L. Exceptions may be considered for patients with ECOG 0-1 who have a history of chronic anemia (80-100 g/L), previous low white blood cell levels (3-4×109/L), or reduced platelets (80-90×109/L). Liver function: ALT and AST <1.5 times the upper limit of normal (ULN), bilirubin <1.5×ULN. Renal function: Serum creatinine (SCR) ≤140 μmol/L.
* Patients are required to provide informed consent to undergo treatment.

Exclusion Criteria:

* Existing or prior history of other malignant tumors (except non-melanoma skin cancer) that are uncontrolled or not cured, depending on the type of the primary tumor.
* Lack of histological or cytological diagnosis for esophageal cancer.
* Previous chest radiotherapy.
* Suffering from innate or acquired immune function defects;
* Pregnancy (confirmed by serum or urine β-HCG test) or during the lactation period; History of drug abuse or alcohol dependence; HIV-positive status, including those on antiretroviral treatment; Chronic hepatitis B with viral replication phase; Active phase of hepatitis C; Active syphilis with a history of mental illness that may hinder treatment completion.
* Poor overall health status, defined as KPS < 70 or ECOG > 2.
* Presence of severe comorbidities that could impact radiotherapy progress, including: Unstable angina, congestive heart failure, or myocardial infarction requiring hospitalization within the past 6 months; Acute bacterial or systemic fungal infections; Exacerbation of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization; Hepatic or renal insufficiency; Immunosuppressed patients; Coexisting connective tissue diseases, such as active scleroderma or lupus, which are contraindications to radiotherapy.
* Inability to comprehend the treatment's purpose or unwillingness to sign the treatment consent form.
* Lack of legal capacity or limited legal capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival | 1 year
  From the initial administration of the study drug to the first identification of disease progression or mortality, whichever happens first. In the case of patients who had not encountered local control failure or death, specifically in terms of progression-free survival, the time of the last tumor assessment was considered as the endpoint. Tumor response was evaluated by investigators following RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Acute toxicity | 3 months
  Monitor the occurrence of acute toxic reactions (based on CTCAE4.03) and subacute toxic reactions (RTOG) in the treatment of cN3 ESCC with the combination of chemotherapy, immunotherapy, and ongoing radiotherapy, both during the treatment course and within three months after its completion.
Quality of Life (QoL) | 1 years
  Collect QoL data on cN3 ESCC patients. The data is measured by EORTC QLQ-C30 (Version 3.0) according to investigator collection at the starting and ending time of the treatment. EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The core and disease-specific for ESCC modules are selected to estimate treatment related influence on patients' life. The final score of the questionnaire is collected and analyzed according to detailed scoring procedures from manuals.
Objective response rate | 1 year
  Defined as the proportion of patients with complete response (CR) or partial response (PR)
Duration of response | 1 year
  Defined as the period from the recognition of an objective response to the first identification of either progression or death, whichever event transpired first.
Disease control rate | 1 year
  Defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD)
Immune Progression Free Survival | 1 year
  defined as the duration from the initial dose of tislelizumab to the first identification of either disease progression or death, whichever happens first. Tumor response was evaluated by investigators following iRECIST criteria.
Overall survival | 1 year
  defined as the period from the initial drug administration to the subject's demise from various causes. In cases where patients were lost to follow-up prior to their passing, the date of their last documented contact was documented. For patients still alive at the last analyzed time point, the time of their last contact was considered as their survival duration. In the analysis of survival and subsequent treatment, all patients were monitored until their death, loss to follow-up, or the conclusion of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No